CLINICAL TRIAL: NCT06775652
Title: Neoadjuvant Chemoradiotherapy Plus Surgery vs. Surgery Plus Adjuvant Therapy for Esophageal Squamous Cell Carcinoma: A Prospective, Randomized Phase III Clinical Trial
Brief Title: Neoadjuvant Chemoradiotherapy Plus Surgery vs. Surgery Plus Adjuvant Therapy for ESCC
Acronym: ESCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, Chief Investigator, Professor of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCH-TS1801
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Esophageal squamous cell carcinoma; Neoadjuvant chemoradiotherapy; Adjuvant therapy; Overall survival; Pathological complete response
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCRT group (Experimental)
  Interventions: Drug: Neoadjuvant Chemoradiotherapy; Procedure: Surgery
- AT group (Active Comparator)
  Interventions: Procedure: Adjuvant therapy; Procedure: Surgery

INTERVENTIONS:
Drug: Neoadjuvant Chemoradiotherapy — Patients assigned to the NCRT group received intravenous paclitaxel (135 mg/m²) and carboplatin (AUC=2-5) on day 1, administered every three weeks for two cycles. Concurrently, they received intensity-modulated radiotherapy (IMRT) with a total of 20 sessions (CTV 40 Gy, GTV 44 Gy) five days per week. All radiotherapy plans were reviewed by designated radiation oncologists before treatment to ensure quality control. Patients were assessed 4 to 6 weeks after completing NCRT following RECIST 1.1 criteria.
  Arms: NCRT group
Procedure: Adjuvant therapy — Patients in the AT group received surgery as soon as possible after randomization, followed by adjuvant therapy, postoperative adjuvant therapy based on pathological staging, as recommended by the NCCN Clinical Practice Guidelines for Esophageal and Esophagogastric Junction Cancers (2017 V4), starting one month post-surgery with either adjuvant chemotherapy or chemoradiotherapy. The adjuvant chemotherapy regimen was the same as the neoadjuvant chemotherapy regimen, and the adjuvant radiotherapy regimen and dose were administered according to guideline recommendations.
  Arms: AT group
Procedure: Surgery — Surgery

SUMMARY:
This phase III randomized clinical trial compared the long-term survival and safety of neoadjuvant chemoradiotherapy (NCRT) followed by surgery versus surgery with adjuvant therapy (AT) in patients with locally advanced esophageal squamous cell carcinoma (ESCC). Conducted at Sichuan Cancer Hospital, patients were randomly assigned to receive either NCRT (chemotherapy and radiotherapy followed by surgery) or AT (surgery followed by adjuvant therapy based on staging).

The primary outcome was overall survival (OS), with secondary outcomes including disease-free survival (DFS), R0 resection rates, and treatment-related toxicity. A total of 245 patients were randomized, and 224 patients were included in the final analysis.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label, phase III clinical trial conducted at Sichuan Cancer Hospital, a high-volume cancer center in China. The primary objective is to compare the long-term survival outcomes of neoadjuvant chemoradiotherapy (NCRT) combined with surgery versus surgery followed by adjuvant therapy (AT) in patients with locally advanced esophageal squamous cell carcinoma (ESCC).

Patients with histologically confirmed, resectable, locally advanced thoracic ESCC (staged according to the 8th edition of the AJCC TNM classification) were enrolled and randomized in a 1:1 ratio to the NCRT or AT group. The NCRT group received intensity-modulated radiotherapy (40 Gy in 20 fractions) combined with paclitaxel and carboplatin, followed by surgery. The AT group underwent surgery first, followed by adjuvant therapy (chemotherapy or chemoradiotherapy) determined by postoperative pathological staging based on the 2018 NCCN Guidelines for Esophageal and Esophagogastric Junction Cancers.

The study's primary endpoint is overall survival (OS). Secondary endpoints include disease-free survival (DFS), R0 resection rate, pathological complete response (pCR) rate, treatment-related toxicity, and postoperative complications. Safety was assessed based on the Common Terminology Criteria for Adverse Events (CTCAE) and the Clavien-Dindo classification for surgical complications.

A total of 245 patients were randomized, with 116 patients in the NCRT group and 108 in the AT group achieving R0 resection and included in the final analysis. Kaplan-Meier survival analysis and Cox proportional hazards models were employed to evaluate OS and DFS.

This trial seeks to provide high-quality evidence for optimizing treatment strategies in locally advanced ESCC and to highlight the significance of achieving pathological response as a predictor of improved survival. Future studies with larger sample sizes and multi-center participation are needed to validate these findings.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 to 75 years, both sexes; 2. Histologically confirmed locally advanced (cT1N+M0 or T2-4aNxM0) thoracic esophageal squamous cell carcinoma (8th UICC-TNM stage); 3. Cervical contrast-enhanced CT showed no suspicious metastatic lymph nodes, and imaging studies confirmed no systemic metastasis; 4. Expected to achieve R0 resection; 5. ECOG performance status 0 to 1; 6. No prior antitumor therapy for esophageal cancer, including chemotherapy, radiotherapy (including planned radiotherapy during the study), hormone therapy, or immunotherapy; 7. Measurable lesions according to RECIST v1.1 criteria; 8. No contraindications for surgery based on preoperative evaluation of organ function; 9. Laboratory test results confirm eligibility:

  * Hemoglobin ≥90 g/L;
  * White blood cell count ≥ the laboratory lower limit of normal;
  * Absolute neutrophil count (ANC) ≥1.5×10⁹/L;
  * Platelet count ≥100×10⁹/L;
  * Total bilirubin ≤1.5× upper limit of normal (ULN);
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN;
  * Prothrombin time ≤16 seconds and international normalized ratio (INR) ≤1.5× ULN;
  * Serum creatinine ≤1.5× ULN or creatinine clearance ≥50 mL/min (calculated using the Cockcroft-Gault formula); 10. Women of childbearing potential must agree to use effective contraception (e.g., intrauterine devices, oral contraceptives, or condoms) during the study medication period and for 60 days after the last dose, have a negative serum pregnancy test within 7 days prior to enrollment, and must not be lactating; 11. Men must agree to use effective contraception during the study medication period and for 60 days after the last dose; 12. Participants must understand and sign the informed consent form.

Exclusion Criteria:

* 1. History of Other Malignancies: 1.1. Patients who have had malignancies other than esophageal cancer.

  2. Bleeding Tendency and Coagulation Disorders: 2.1. Gastrointestinal bleeding within 6 months prior to randomization. 2.2. Coagulation disorders at the time of enrollment. 2.3. Patients receiving thrombolysis or anticoagulant therapy.

  3. Cardiovascular and Cerebrovascular Diseases: 3.1. The following conditions within 12 months prior to randomization:
  * Congestive heart failure classified as NYHA class II or higher.
  * Unstable angina, myocardial infarction, or poorly controlled arrhythmias.
  * Cerebrovascular accidents. 3.2. Left ventricular ejection fraction (LVEF) <50% on echocardiography. 3.3. Corrected QT interval (QTc) >480 ms (calculated using the Fridericia formula; if QTc is abnormal, three consecutive tests should be conducted at 2-minute intervals, and the average value used).

3.4. Medically difficult-to-control hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg) based on the average of at least two measurements.

3.5. History of hypertensive crises or hypertensive encephalopathy.

4. Respiratory Diseases: 4.1. History of interstitial lung disease or pneumonia requiring steroid treatment at enrollment.

4.2. Active tuberculosis at the time of randomization or anti-tuberculosis treatment within 1 year prior to randomization.

4.3. Asthma requiring intermittent bronchodilators or other medical interventions at randomization.

5. Infectious and Inflammatory Diseases: 5.1. Patients with active hepatitis B must receive effective treatment before enrollment.

5.2. For patients positive for HCV antibodies, HCV-RNA testing should exclude those with HCV-RNA >10³ copies/mL.

5.3. Co-infection with HIV.

6. Surgery-Related Risks: 6.1. Severe unhealed wounds, active ulcers, or untreated fractures at the time of randomization.

6.2. Other conditions rendering the patient inoperable. 6.3. Prior surgeries that preclude using the stomach for esophageal reconstruction during this surgery.

7. Drug and Treatment-Related Risks: 7.1. Receiving systemic steroid therapy (daily prednisone >10 mg or equivalent) or other immunosuppressive agents within 2 weeks before randomization.

7.2. Severe allergy to chemotherapy drugs. 7.3. Previous organ transplant recipients.

8. Liver Function Requirements: 8.1. For patients with HBsAg(+) and/or HBcAb(+), HBV DNA must be <500 IU/mL with normal liver function.

8.2. Continued effective anti-HBV therapy during the study or initiation of entecavir or tenofovir treatment prior to study medication.

9. Other Conditions: 9.1. Severe unhealed wounds, active ulcers, or untreated fractures at the time of randomization.

9.2. Any condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
OS | 5 years
  Overall survival

SECONDARY OUTCOMES:
DFS | 5 years
  Disease-free survival
Adverse Events | 1 years
  Treatment-related toxicity, postoperative complications
R0 resection rate | 1 years
  Other outcomes
pathological complete response (pCR) rate | 1 years
  Other outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
This study aims to compare the long-term survival outcomes and safety profiles of neoadjuvant chemoradiotherapy (NCRT) followed by surgery versus surgery with adjuvant therapy (AT) in patients with locally advanced esophageal squamous cell carcinoma (ESCC). The study follows a prospective, randomized, open-label, phase III clinical trial design. Eligible patients were assigned in a 1:1 ratio to receive either NCRT followed by surgery or surgery with AT, with treatment assignments stratified by a permuted-block randomization method. Key endpoints include overall survival (OS), disease-free survival (DFS), pathological outcomes, and treatment-related adverse events. This research emphasizes the importance of pathological complete response (pCR) as a predictor of improved survival and aims to provide robust evidence to guide treatment strategies for locally advanced ESCC. Data collection, patient follow-up, and statistical analyses were conducted in accordance with international clinical
Supporting Information: Study Protocol

REFERENCES:
- [Derived] He W, Li Z, Xie Q, Han Y, Peng L, Wang C, Wang K, Liu G, Li H, Zhou Q, Li J, Zhang H, Xiao W, Fang Q, Miao Y, Leng X. Long-Term Survival Outcomes of NCRT With Surgery vs Surgery With Adjuvant Therapy for ESCC: A Single-Center Prospective Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2550307. doi: 10.1001/jamanetworkopen.2025.50307. PMID 41490111